CLINICAL TRIAL: NCT01909817
Title: A Novel Method for Enhancement of Standard Rest Electrocardiograms (ECG) Provides New Parameters for Early Detection of Coronary Artery Disease (CAD)
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: HYMC-9-2003
Record Dates: First submitted 2013-03-20; First posted 2013-07-29 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2013-07

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Routine coronary angiogram patients
  Interventions: Procedure: Routine coronary angiogram

INTERVENTIONS:
Procedure: Routine coronary angiogram

SUMMARY:
The investigators aim to determine whether a new method of enhancing and improving ECG acquisition, analysis and display is effective. The investigators will perform superimposition and summation of multiple standard ECG cycles, in the same lead, by temporal alignment to the peak R wave and voltage alignment to an improved baseline at the T-P segment.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing routine coronary angiogram

Exclusion Criteria:

* Patients with significant irregular heart rhythm
* Patients with heart failure

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing routine coronary angiogram
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2013-07; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
ECG Voltage spread | One month
  We will measure the voltage spread at the S-T and P-R intervals after superimposition and summation of multiple standard ECG cycles in the same lead, by temporal alignment to the peak R wave and voltage alignment to an improved baseline at the T-P segment.

CONTACTS AND LOCATIONS:
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel